CLINICAL TRIAL: NCT02842892
Title: Implication of Stiffness of the Hamstrings, Achilles Tendon and Calf Muscles for Jumping Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Winfried Banzer, Head of Department, Goethe University
Purpose: Diagnostic
Other Study IDs: SpM2016-004
Record Dates: First submitted 2016-07-18; First posted 2016-07-25 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Tissue Compliance

ARMS (3):
- Squat Jump (Other)
  Interventions: Other: Tissue stiffness
- Drop Jump (Other)
  Interventions: Other: Tissue stiffness
- Countermovement Jump (Other)
  Interventions: Other: Tissue stiffness

INTERVENTIONS:
Other: Tissue stiffness

SUMMARY:
For optimal jumping performance an adequate interaction of muscles and tendons is required. A parameter in the functional evaluation of both structures is their stiffness (resistance of the tissue against deformation by external forces). It is unclear so far if higher stiffness values of tendon or muscle or a specific stiffness relation of both tissues is the cause of better jumping performance. The present study examines this based on the Achilles tendon and the calf muscles or the patellar tendon and the hamstrings by three different forms of jumps (squat jump, counter-Movement Jump, Drop-Jump).

The plan is to include young healthy volunteers aged 18 to 40 years. In a cross-sectional study, the jump height of the participants will be measured for each jump form: squat jump (jump from a squatting position), Counter-Movement Jump (jump with backswing by going into the knees) or drop jump (jump from small box with direct re-jump). The order of the jump form is determined randomly. The measurements are carried out within one day. Furthermore the international physical activity questionnaire will be used in order to assess the level of physical activity.

As primary outcome the stiffness of the calf muscles, achilles tendon, hamstring and patellar tendon will be detected. The measurement is carried out before the jumps (there are three jumps after one sample jump performed). The measurement is executed non-invasively and completely painless using Indentometers and MyotonPro. With both devices, minimal pressure on the examined tissue will be exerted and measured how much of this can be compressed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Drug intake in the past 48 hours
* Pregnancy
* Muscle soreness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Tissue Stiffness (calf muscles, achilles tendon, hamstring and patellar tendon) using two different tissue compliance meter (Indentometer Pro; Myoton Pro). | 15 Min.

SECONDARY OUTCOMES:
Jumping performance (counter movement jump, drop jump, squat jump) using a contact time mat (Refitronic) | 10 Min

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sports Medicine, Goethe University Frankfurt/Main, Frankfurt am Main, Hesse, Germany